CLINICAL TRIAL: NCT07375277
Title: Effects Of Biceps Transposition Without Tenotomy For Augmentation Of Massive Rotator Cuff Repairs On Function, Quality Of Life, And Sleep: A Prospective Study
Brief Title: Effects Of Biceps Transposition Without Tenotomy For Augmentation Of Massive Rotator Cuff Repairs
Acronym: ROTATORCUFF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, güneş sarıkaya, BALIKESİR CİTY HOSPİTAL, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCH-BTA-MRCR-2026-001
Record Dates: First submitted 2026-01-17; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Massive Rotator Cuff Tear
Keywords: Biceps Transposition; Massive Rotator Cuff Tear; Arthroscopic Partial Repair

STUDY DESIGN:
Intervention Model Description: Single-arm, single-group study in which all participants undergo arthroscopic partial rotator cuff repair augmented with tenotomy-sparing long head of the biceps tendon (LHBT) transposition, with outcomes assessed at baseline, 3 months, and 12 months.
Masking Description: This is an open-label, single-arm interventional study. Due to the nature of the surgical intervention, participants, care providers, investigators, and outcome assessors are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biceps Transposition Augmentation (Other): Participants in this single arm undergo arthroscopic partial rotator cuff repair augmented with tenotomy-sparing transposition of the long head of the biceps tendon (LHBT). All procedures are performed according to a standardized surgical and rehabilitation protocol.
  Interventions: Procedure: LHBT Transposition Augmentation

INTERVENTIONS:
Procedure: LHBT Transposition Augmentation — Arthroscopic partial rotator cuff repair augmented with transposition of the intact long head of the biceps tendon (LHBT) without tenotomy. The transverse humeral ligament is released to mobilize the tendon, which is transposed and fixed to the greater tuberosity footprint using a standardized anchor/suture technique to support the partial repair. Procedures are performed under a standardized surgical and postoperative rehabilitation protocol.

SUMMARY:
This prospective, single-arm interventional study will evaluate the effects of long head of the biceps tendon (LHBT) transposition without tenotomy as an augmentation technique for arthroscopic partial repair in adults with massive rotator cuff tears. Consecutive eligible patients undergoing arthroscopic partial rotator cuff repair plus tenotomy-sparing LHBT transposition augmentation at Balikesir City Hospital (Balikesir, Turkiye) will be enrolled and followed for 12 months. Patient-reported outcomes and clinical assessments will be collected preoperatively (baseline) and postoperatively at 3 and 12 months. The primary outcomes are shoulder function (ASES), rotator cuff-related quality of life (WORC converted to a 0-100 scale), and sleep disturbance (Insomnia Severity Index). Secondary outcomes include active shoulder range of motion and biceps-related clinical findings (Speed test, Yergason test, bicipital groove tenderness, and Popeye deformity). Postoperative MRI will not be obtained routinely and will be performed only if clinically indicated. The study aims to provide standardized prospective data on functional outcomes, quality of life, and sleep after this augmentation approach.

DETAILED DESCRIPTION:
Detailed Description Massive rotator cuff tears may not be amenable to full anatomic repair, and even when partial repair is feasible, residual symptoms and functional limitations may persist. Long head of the biceps tendon (LHBT) transposition without tenotomy has been proposed as an augmentation strategy that may provide additional biomechanical and biologic support to arthroscopic partial rotator cuff repair. However, prospective data with standardized follow-up evaluating functional outcomes, rotator cuff-specific quality of life, and sleep outcomes remain limited. This study is designed to generate prospective, standardized clinical and patient-reported outcome data after tenotomy-sparing LHBT transposition augmentation in the setting of massive rotator cuff repair.

This is a prospective, single-arm, non-randomized interventional clinical study conducted at Balikesir City Hospital, Department of Orthopedics and Traumatology (Balikesir, Turkiye). Consecutive eligible adult patients will be enrolled between January 2026 and December 2026, with a planned sample size of 35 participants. Each participant will be followed for a minimum of 12 months. Assessments will be performed preoperatively (baseline) and postoperatively at 3 months and 12 months.

Participants and Eligibility Massive rotator cuff tear will be defined on preoperative MRI as a full-thickness tear involving at least two tendons and/or a tear with the greatest dimension greater than 5 cm. Final eligibility will be confirmed intraoperatively when the tear pattern is deemed suitable for arthroscopic partial repair with LHBT augmentation. Inclusion criteria include age 18 years or older, persistence of symptoms despite at least 3 months of standard nonoperative treatment, planned arthroscopic partial repair with LHBT augmentation, intact LHBT at the time of surgery, and willingness to attend the scheduled follow-up visits. Exclusion criteria include tear patterns not requiring augmentation (e.g., preserved rotator cable patterns), conditions affecting shoulder function (e.g., relevant neurologic disease, inflammatory arthritis), active infection, systemic conditions preventing protocol rehabilitation, inability to provide informed consent, or expected nonadherence to follow-up.

Intervention and Standardization All surgeries will be performed arthroscopically under general anesthesia (with or without interscalene block per anesthesia protocol) in the beach-chair position. Standard diagnostic glenohumeral assessment and subacromial bursectomy will be performed. Acromioplasty may be performed routinely per the surgical standard. The rotator cuff will be mobilized and partially repaired to achieve acceptable tension. For augmentation, the LHBT will be confirmed intact and will not be tenotomized. The transverse humeral ligament will be released to mobilize the tendon. The tendon will be transposed posterior to the bicipital groove and directed to the superior aspect of the greater tuberosity, avoiding overtension. Fixation will be performed to the footprint region using a standardized anchor/suture technique to create an augmentation construct supporting the partial repair. Arthroscopic assessment will confirm absence of overtension and mechanical impingement. Concomitant procedures (e.g., subscapularis repair, distal clavicle resection) will be performed only when clinically indicated and will be recorded.

Rehabilitation Protocol Postoperative management will be standardized: sling immobilization for 3 weeks; passive range of motion initiated immediately in the early postoperative period within pain limits; active range of motion starting at postoperative week 4; strengthening at approximately postoperative month 3. Biceps loading will be restricted for the first 4 weeks (no resisted elbow flexion or supination), followed by gradual progression. Rehabilitation adherence and protocol deviations will be documented.

Imaging and Intraoperative Measurements Preoperative MRI will be evaluated using the Patte classification (retraction) and Goutallier grading (fatty degeneration) by two independent assessors, with disagreements resolved by consensus. Preoperative radiographs will include Hamada classification and acromiohumeral interval (mm). Intraoperatively, tear dimensions (anteroposterior and mediolateral) will be measured using a calibrated probe at the footprint level; tear area will be recorded using a standardized practical approach (e.g., AP × ML). Routine postoperative MRI will not be performed and will be obtained only if clinically indicated (e.g., sudden strength loss, trauma, suspected failure).

Outcomes Primary outcomes are changes in ASES score, WORC score (reported on a 0-100 scale), and Insomnia Severity Index (ISI) from baseline to 3 and 12 months. WORC will be converted to a 0-100 scale using the formula: WORC (0-100) = [1 - (raw WORC / 2100)] × 100, where higher scores indicate better status. Secondary outcomes include active shoulder range of motion (forward elevation, abduction, external rotation by goniometer; internal rotation recorded using a standard method) and biceps-related clinical findings (Speed test, Yergason test, bicipital groove tenderness, Popeye deformity) assessed at baseline, 3 months, and 12 months.

Safety, Data Management, and Analysis All adverse events and complications will be recorded throughout follow-up, and clinically indicated standard care will be provided when needed. Participant data will be de-identified using unique study IDs and stored in password-protected, access-restricted electronic files. Data quality will be supported by random source verification of approximately 10% of records. Statistical analyses will use two-sided significance level of p < 0.05. Longitudinal changes across time points (baseline, 3 months, 12 months) will be analyzed using linear mixed-effects models (time as fixed effect; participant as random intercept), with appropriate adjustment for multiple comparisons (e.g., Holm-Bonferroni). If assumptions are violated, nonparametric repeated-measures methods will be used as sensitivity analyses. Binary outcomes will be analyzed using appropriate paired/repeated methods (e.g., McNemar for two time points; mixed-effects logistic regression for three time points). Effect sizes and 95% confidence intervals will be reported, and missing data patterns will be described with complete-case sensitivity analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of a massive rotator cuff tear on preoperative MRI, defined as a full-thickness tear involving at least two tendons and/or a tear with a greatest dimension greater than 5 cm
* Planned arthroscopic partial rotator cuff repair with augmentation using tenotomy-sparing long head of the biceps tendon (LHBT) transposition
* Persistence of symptoms despite at least 3 months of standard nonoperative treatment
* Intact LHBT confirmed intraoperatively
* Willingness and ability to attend scheduled follow-up visits (baseline, 3 months, and 12 months)
* Provision of written informed consent

Exclusion Criteria:

Exclusion Criteria:

* Tear patterns not requiring augmentation (e.g., preserved rotator cable patterns)
* Neurologic conditions, inflammatory arthritis, active infection, or systemic conditions that may affect shoulder function or prevent protocol rehabilitation
* Inability to provide informed consent
* Expected nonadherence to follow-up or rehabilitation protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Score | aseline, 3 months, and 12 months postoperatively
  The ASES score is a validated patient-reported outcome measure assessing shoulder pain and function on a 0-100 scale, with higher scores indicating better shoulder function.

CONTACTS AND LOCATIONS:
Overall Officials: özgün 0 karakuş, M.D, Study Director — Balikesir Ataturk City Hospital
Locations (1):
- Güneş Sarıkaya, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No